CLINICAL TRIAL: NCT03199066
Title: The Incidence, Epidemiology, Clinical Characteristic, Prognostic Factors, Therapy and Outcome of Non-Hodgkin Lymphoma Patients in the Czech Republic. NiHiL- Longitudinal Observational Study of Czech Lymphoma Study Group (CLSG)
Brief Title: Non-Hodgkin Lymphoma - Observational Epidemiological and Clinical Study (NiHiL)
Status: Recruiting | Type: Observational
Sponsor: Czech Lymphoma Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: NiHiL
Record Dates: First submitted 2017-06-14; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Non Hodgkin Lymphoma (NHL)
Keywords: survival; therapy; epidemiology
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- All NHL subtypes: no interventions
- DLBCL: only patients with diffuse large B-cell lymphoma
- FL: only patients with follicular lymphoma
- MCL: only patients with mantle cell lymphoma
- SLL/CLL: only patients with small lymphocytic lymphoma / chronic lymphocytic leukemia
- MZL: only patients with marginal zone lymphoma
- other B-cell lymphomas: only patients with B-lymphomas not described above
- T-cell lymphomas: only patients with all types of T-cell lymphoma

SUMMARY:
The Czech National Lymphoma Registry (NiHiL) was founded to monitor epidemiologic data and improve the diagnostic evaluation and quality of treatment of patients with non-Hodgkin´s lymphoma (NHL).

The patients are registered into the registry in anonymized form. For each patient are available: registration form, diagnostic form, treatment form, follow- up form, and other malignancy form.

Data quality in the NiHiL has been checked by audits. The data is analyzed according to NHL subtypes with endpoints: lymphoma distribution, epidemiological data, prognostic characteristic, treatment characteristics, response rate, relapse rate, mortality, PFS, OS, DFS, Lymphoma specific survival, longterm toxicity.

DETAILED DESCRIPTION:
The Czech National Lymphoma Registry (NiHiL) was established in 1999 in order to monitor epidemiologic data and to improve the diagnostic evaluation and quality of treatment of patients with non-Hodgkin´s lymphoma (NHL). The database NiHiL includes majority of patients with NHL in the Czech Republic, treated in one of seven University Hospitals and other smaller centres. This represents approx. 75% of all lymphoma patients in the Czech Republic. Since 1999 until the end of year 2016 there were registered 14000 pts.

The patients are registered into the registry in anonymized form at the time of diagnosis after signing informed consent and data are updated/collected at the end of first line treatment, at each relapse including therapy for relapse and then annual follow-up and at the time of death. The registration is submitted electronically via secure internet system. For each patient are available following forms: registration form, diagnostic form, treatment form, follow- up form, and other malignancy form. The content of diagnostic form consists of diagnosis according WHO classification including the copy of original histology description, date of diagnosis, clinical stage, B symptoms, nodal and extranodal involvement, laboratory findings and prognostic systems (IPI, aaIPI, MIPI, FLIPII and others). The prognostic system is calculated automatically. The diagnostic form is the same for the first diagnosis and for the relapses. The treatment form consists of detailed information on the treatment: chemotherapy regimens, therapy with monoclonal antibodies, radiotherapy, autologous or allogeneic transplant. Response assessment has been adjusted to the different version of Chesson criteria for malignant lymphoma. It is expected that comorbidity score and toxicities evaluation will be added into the therapeutic form too.

The follow-up form is requested to be updated annually, besides that in case of relapse or death. This form includes information about clinical status, date of relapse or death.

The exports made from NiHiL content all data from registry and survival data (overall survival, progression survival and disease free survival).

Data quality in the NiHiL has been checked by audits recently, which have been carried out in each centre twice a year.

The data is analyzed according to NHL subtypes with endpoints: lymphoma distribution, epidemiological data, prognostic characteristic, treatment characteristics, response rate, relapse rate, mortality, PFS, OS, DFS, Lymphoma specific survival, longterm toxicity.

The registry has been repeatedly supported by the grants of Ministry of Health. A substantial number of papers originated from the NiHiL have been published in last 15 years in both Czech and international journals. The main aim of the registry is to collect data for malignant lymphoma for better understanding of epidemiological and clinical data about this disease.

ELIGIBILITY:
Inclusion Criteria:

* lymphoma diagnosis
* treated in the Czech Republic
* signed informed consent

Exclusion Criteria:

* unsigned informed consent
* age <18 y

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: new patients with non-Hodgkin´s lymphoma (NHL)
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 1999-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
lymphoma epidemiology in CZ | On average once a year
  occurrence and study of factors influencing the formation of non-hodgkin´s lymphoma from data filled into registry forms by physicians and datamangers

SECONDARY OUTCOMES:
clinical characteristics | On average once a year
  patients clinical characteristics from data filled into registry forms by physicians and datamangers (values of lactate dehydrogenase, clinical stage, performance status, age ≥ 60 years and number of extranodal localizations will be combined to report IPI /International prognostic index/; other prognostic risk factors will be calculated similarly)
biological characteristics | On average once a year
  patients biological characteristics from data filled into registry forms by physicians and datamangers (immunohistochemical differences of non-hodgkin´s lymphomas, e.g. GC-like or non GC-like phenotype of DLBCL)
prognostic systems | On average once a year
  evaluation of prognostic factors based on subtypes of lymphoma from data filled into registry forms by physicians and datamangers
therapy used | On average once a year
  type of therapy - induction or following therapy - for all patients from data filled into registry forms by physicians and datamangers
patients outcome | On average once a year
  Overall response is measured according to Revised Response Criteria For Malignant Lymphoma (Cheson BD et al, JCO 2007; the main examinations PET/CT and bone marrow biopsy) for all patients, who can be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Marek Trneny, prof. MD, Principal Investigator — Charles University General Hospital, Prague, CZ
Locations (1):
- Charles University General Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data are available only for reasearchers in CLSG.

REFERENCES:
- [Derived] Vodicka P, Janikova A, Belada D, Hanackova V, Mocikova H, Duras J, Steinerova K, Benesova K, Konirova E, Prochazka T, Polgarova K, Masar M, Dlouha J, Blahovcova P, Trneny M. Long-Term Real-World Outcomes of Primary CNS Lymphoma Patients Treated With MATRix Regimen Are Similar to IELSG32 Trial Results. Hematol Oncol. 2025 Nov;43(6):e70142. doi: 10.1002/hon.70142. PMID 41108618
- [Derived] Mocikova H, Pytlik R, Benesova K, Janikova A, Duras J, Sykorova A, Steinerova K, Prochazka V, Campr V, Belada D, Trneny M. Peripheral T-Cell Lymphomas Involving the Central Nervous System: A Report From the Czech Lymphoma Study Group Registry. Front Oncol. 2022 May 12;12:874462. doi: 10.3389/fonc.2022.874462. eCollection 2022. PMID 35646641
- [Derived] Vodicka P, Benesova K, Janikova A, Prochazka V, Belada D, Mocikova H, Steinerova K, Duras J, Karban J, Hanackova V, Sykorova A, Obr A, Trneny M. Polatuzumab vedotin plus bendamustine and rituximab in patients with relapsed/refractory diffuse large B-cell lymphoma in the real world. Eur J Haematol. 2022 Aug;109(2):162-165. doi: 10.1111/ejh.13784. Epub 2022 May 11. PMID 35502609
- [Derived] Lobello C, Tichy B, Bystry V, Radova L, Filip D, Mraz M, Montes-Mojarro IA, Prokoph N, Larose H, Liang HC, Sharma GG, Mologni L, Belada D, Kamaradova K, Fend F, Gambacorti-Passerini C, Merkel O, Turner SD, Janikova A, Pospisilova S. STAT3 and TP53 mutations associate with poor prognosis in anaplastic large cell lymphoma. Leukemia. 2021 May;35(5):1500-1505. doi: 10.1038/s41375-020-01093-1. Epub 2020 Nov 27. No abstract available. PMID 33247178
- See also: Official Site of the Czech Lymphoma Study Group — https://www.lymphoma.cz/studies/kls_nihil.php